CLINICAL TRIAL: NCT05683483
Title: WEsleep Trial: Improving Sleep With Non-pharmalogical Interventions in Hospitalized Patients
Brief Title: WEsleep Trial: Improving Sleep in Hospitalized Patients
Acronym: WEsleep
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Dirk Jan Stenvers, Endocrinologist, Principal Investigator, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: WEsleep Trial
Record Dates: First submitted 2022-12-23; First posted 2023-01-13 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Sleep; Sleep Disturbance; Sleep Hygiene; Circadian Dysrhythmia; Surgery; Sleep Disorders, Circadian Rhythm
MeSH Terms: conditions — Parasomnias; Sleep Hygiene; Sleep Disorders, Circadian Rhythm

STUDY DESIGN:
Intervention Model Description: We will perform a cluster randomized controlled trial. Randomization will be stratified, to ensure that departments are comparable at baseline in terms of types of patients, and that not all intervention departments are in one of our two locations and all control departments in the other location..
Masking Description: As interventions will be implemented on the level of the department (for 6 departments), it will not be possible to blind health care providers, researchers or patients for the intervention that the patient is receiving.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Surgical WEsleep (Experimental): Patients admitted into the 3 surgical departments/clusters where the WEsleep interventions are implemented.
  Interventions: Other: WEsleep Interventions
- Medical WEsleep (Experimental): Patients admitted into the 3 non-surgical departments/clusters where the WEsleep interventions are implemented
  Interventions: Other: WEsleep Interventions
- Surgical Standardcare (No Intervention): Patients admitted into the 3 surgical departments/clusters where the WEsleep interventions are NOT implemented, and patients are receiving standardcare
- Medical Standardcare (No Intervention): Patients admitted into the 3 non-surgical departments/clusters where the WEsleep interventions are NOT implemented, and patients are receiving standardcare

INTERVENTIONS:
Other: WEsleep Interventions — 1) Postponing morning nursing rounds to avoid waking patients early and daily assessment of sleep quality by the nurse during morning rounds; 2) Implementing sleep promoting interventions, including optimization of medication and iv fluid timing; 3) Education for health care professionals on sleep; 4) Implementing sleep rounds and change department infrastructure; including 'sleep menu' where patients can choose from earplugs, eye masks, and warm socks. Implement blackout curtains depending on baseline light intensity.
  Arms: Medical WEsleep; Surgical WEsleep

SUMMARY:
In the WEsleep study, the investigators will perform a cluster randomized controlled trial. 3 surgical and 3 medical departments will be randomized to implement low-cost and simple interventions aimed at improving sleep in admitted patients. Another 3 surgical and 3 medical departments will be randomized to function as control groups. Subjective sleep quality and sleep-wake timing will be assessed in adult medical and surgical patients admitted into one of 12 participating wards, using questionnaires and a sleep diary. In addition, in a subset of participants, objective sleep measures will be assessed in with an EEG headband and a sleep mat.

DETAILED DESCRIPTION:
Objectives

Primary objective

Our primary objective is to investigate whether a set of low-cost and easily applicable interventions improves subjective sleep quality of hospitalized patients on the second night of admission (for medical patients) and first postoperative night (for surgical patients) as measured the Richards-Campbell sleep questionnaire, comparing between intervention and control departments.

Secondary objectives

* To investigate whether the WEsleep interventions improves subjective sleep quality for all night of admission (max. 7)
* To investigate whether the WEsleep interventions reduced the lowering of subjective sleep quality during admission when compared to subjective sleep quality before admission (on a work-free day 30 days before admission, retrospectively assessed at inclusion)
* To investigate whether the disruption of the circadian timing system (as measured by the diurnal phase shift of midpoint of sleep) was smaller for patients in the intervention group on the first postoperative night for surgical patients and the second night of admission for medical patients
* To investigate whether the WEsleep interventions reduced night-to-night changes in subjective sleep-wake timing (i.e. midpoint of sleep, on- and offset, duration, latency, inertia and daytime napping) for all nights of admission (max. 7)
* To investigate the association between the timing of food intake (i.e. first and last meal of the day and whether food was eaten after 21:00h) and sleep quality and timing.
* To investigate the association between quality of recovery and sleep quality and sleep-wake timing
* To investigate 30-day mortality for patients admitted into intervention and control departments
* To investigate 30-day incidence of delirium for patients admitted into intervention and control departments
* For surgical patients: to investigate the 30-day incidence of surgical site infections
* Objective sleep substudy: to investigate the difference between intervention and control departments in objective sleep efficiency of hospitalized patients on the second night of admission (in medical patients) and the first postoperative night on ward (in surgical patients) as measured by the Dreem-3 EEG-headband
* Objective sleep substudy: to investigate whether the WEsleep interventions reduced night-to-night changes in objective sleep-wake timing (i.e. midpoint of sleep, on- and offset, duration, latency, inertia and daytime napping) for all nights of admission (max. 7)
* Objective sleep substudy: to investigate whether the WEsleep interventions influence night-to-night changes in objective sleep measures (as measured by the Dreem 3 EEG-headband and Withings Sleep analyzer) for all nights of admission (max. 7)
* Objective sleep substudy: to investigate the difference between objective sleep measures (as measured by Dreem-3 EEG-headband and Withings Sleep Analyzer) and subjective sleep measures (as measured by the Richard Campbell Sleep Questionnaire and the Consensus Sleep Diary) for a population of hospitalized medical and surgical patients
* Objective sleep substudy: to investigate the association between quality of recovery and objective sleep quality and sleep-wake timing
* Objective sleep substudy: to investigate the association between 30-day mortality and objective sleep quality and quantity
* Objective sleep substudy: to investigate the association between 30-day incidence of delirium and objective sleep quality and quantity
* Objective sleep substudy: to investigate the association between the 30-day incidence of surgical site infections and objective sleep quality and quantity (for surgical patients)

Study Procedure:

6 departments will be randomized (3 surgical, 3 medical) to receive the WEsleep-interventions, which will consist of: 1) Postponing morning nursing rounds to avoid waking patients early and daily assessment of sleep quality by the nurse during morning rounds; 2) Implementing sleep promoting interventions, including optimization of medication and iv fluid timing; 3) Education for health care professionals on sleep; 4) Implementing sleep rounds and change department infrastructure; including 'sleep menu' where patients can choose from earplugs, eye masks, and warm socks. Implement blackout curtains depending on baseline light intensity.

Implementation of the interventions will be evaluated on a regular basis throughout the length of the study to make sure that all interventions are provided to our patients as planned.

Before implementation, a baseline measurement will be conducted on all participating departments in a small number of patients (which is not part of the sample size). After study onset, we observed that some interventions were gradually implemented. As such, we decided that for optimal assessment of the effect of the intervention a run-in period of 12 weeks before starting assessment of the primary and secondary outcomes would be reasonable. Sleep measurements between study onset and outcome will be used to guide implementation and will be reported in eventual journal articles. After 12 weeks (that is, after July 1st), 33 patients per participating department will be included, for a total of 396 patients (12 departments with 33 patients each) and analyzed for the outcomes of the study. Informed consent for sleep measurements will be obtained on the first or second day of admission into one of the participating wards. Patients will be followed until discharge or for a maximum of 7 nights of admission. Patient characteristics, as well as data on the admission will be extracted from the electronic medical record.

In the objective sleep substudy, 24 patients will be recruited from each group (medical intervention and control groups, surgical intervention and control groups), for a total of 96 patients. Measurements between April 11th and June 30th will be used to guide implementation of interventionsPatients included after July 1st will be analyzed for the outcomes of the substudy. Informed consent for the substudy will be obtained separately at the same time as consent for the main study. All patients participating in the main study will be asked to participate in the substudy as well. After obtaining consent, a lottery system will decide which patients can participate in the substudy (due to the scarcity of available Dreem-3 EEG headbands and Withings Sleep Analyzers). Patients will be asked to complete two questionnaires daily:

Richards Campbell Sleep Questionnaire (RCSQ) on subjective sleep quality Consensus Sleep Diary (CSD) for day-to-day sleep wake timing during admission Furthermore, patients are asked at admission to complete the two questionnaires on sleep quality and sleep-wake timing on work- and work-free days (RCSQ and CSD) retrospectively, i.e. for 30 days before admission. Patients will also complete a Quality of Recovery 15 (QoR-15) questionnaire twice (once at one day after surgery/first day of admission and once three days after surgery/third day of admission).

In the substudy, objective sleep in patients will be measured with the Dreem-3 EEG-headband and the Withings Sleep Analyzer. The Dreem-3 headband uses electro-encephalography (EEG) and a validated algorithm to differentiate between wakefulness and various sleep stages (Rapid-Eye Movement (REM)-sleep and non-REM N1, N2 and N3 sleep) and the time at which these occur. The Withings Sleep Analyzer can be placed under the mattress and uses measurement of movement to differentiate between wakefulness and light, deep and REM-sleep and the times at which these occur.

ELIGIBILITY:
Surgical: Patients admitted for elective surgery with planned overnight stay Medical:Patients admitted to the medical ward, with at least two expected nights of admission

Inclusion Criteria:

Surgical patients:

* Adult (18+) patients
* Undergoing elective non-cardiac surgery with planned (post-operative) overnight stay
* Willing and able to provide informed consent
* Able to read and write in Dutch

Medical patients:

* Adult (18+) patients medical admission with expected stay of at least two nights
* Willing and able to provide informed consent
* Able to read and write in Dutch

Exclusion Criteria:

* Surgical patients: ASA score of 4 or higher
* Surgical patients: PACU admission during first postoperative night
* Admission on ICU-ward at any time during admission (both planned and unplanned, for both surgical and medical patients)
* Non-Dutch speaking
* Strict isolation (MRSA or aerogenic isolation)
* Pre-existing delirium or cognitive impairment

NB: After starting inclusions, some patients were found to spend the first postoperative night on post-anesthesia care unit (PACU) instead of a WEsleep intervention or control department and after deliberation this was added as a criterium for exclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 396 (Actual)
Dates: Start 2023-04-11 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
Subjective Sleep Quality during admission | Second night of admission (for medical patients), first postoperative night on ward (for surgical patients)
  Subjective sleep quality will be assessed with the Richard Campbell Sleep Questionnaire (RCSQ). The RCSQ measures sleep quality on five questions using a visual analogue scale (VAS), ranging from 0 to 100, with higher scores indicating a better sleep quality.
  A sixth question was added to assess noise levels (as is quite customary), using a VAS-scale, ranging from 0-100, with a higher score indicating more noise

SECONDARY OUTCOMES:
Night-to night changes in subjective sleep quality | The first night until the seventh night of admission; if the patient is discharged before 7 nights of admission, all nights of admission will be analyzed
  Subjective sleep quality will be assessed with the Richard Campbell Sleep Questionnaire (RCSQ). The RCSQ measures sleep quality on five questions using a visual analogue scale (VAS), ranging from 0 to 100, with higher scores indicating a better sleep quality.
  A sixth question was added to assess noise levels (as is quite customary), using a VAS-scale, ranging from 0-100, with a higher score indicating more noise
Difference in subjective sleep quality between during admission and at home | Second night of admission vs. a work- and workfree day 30 days before admission
  Subjective sleep quality will be assessed with the Richard Campbell Sleep Questionnaire, with five questions on a visual analogue scale, ranging from 0 to 100, with higher scores indicating better sleep quality. For this outcome, we will assess the subjective sleep quality at home retrospectively at inclusion.
Diurnal phase shift of sleep-wake timing | Second night of admission (for medical patients) or first postoperative night (for surgical patients) vs. a workfree day 30 days before admission
  The phase shift of sleep-wake timing will be assessed by comparing midpoint of sleep during admission with midpoint of sleep on a work-free day before admission, both measured with the Consensus Sleep Diary (CSD). For this outcome, we will assess sleep-wake timing at home retrospectively at inclusion.
Night-to-night changes in sleep-wake timing | The first night until the seventh night of admission; if the patient is discharged before 7 nights of admission, all nights of admission will be analyzed
  The changes in sleep-wake timing (i.e. midpoint of sleep, sleep on- and offset time, sleep duration, sleep latency & inertia and daytime napping), as measured by the CSD.
Timing of food intake and sleep quality/timing | The first night until the seventh night of admission; if the patient is discharged before 7 nights of admission, all nights of admission will be analyzed
  The association between food intake timing (i.e. first and last meal of the day and whether food was eaten after 21:00h), as measured by asking patients directly for the time of the first and last meal of the day and whether patients ate after 21:00h), and subjective sleep quality and sleep-wake timing (as measured by the Richard Campbell Sleep Questionnaire (with five questions on a visual analogue scale ranging from 0-100 with higher scores indicating better sleep quality) and Consensus Sleep Diary (with questions on sleep-wake timing) respectively).
Quality of recovery (for surgical patients) and sleep quality/timing | First and third day after surgery
  The association between quality of recovery (in surgical patients), as measured by the Quality-of-Recovery 15 item questionnaire (QoR-15), and subjective sleep quality and sleep-wake timing (as measured by the Richard Campbell Sleep Questionnaire and Consensus Sleep Diary respectively). The QoR-15 will be completed twice by patients.
30 day mortality | 30 days after admission
  30-day mortality, assessed by checking the medical record retrospectively 30 days after admission.
30-day incidence of delirium during admission | 30 days after admission
  30-day incidence of the clinical diagnosis of delirium during hospitalization, as assessed by a physician during admission. Patients will be assessed for delirium at the request of nursing staff or if the score of the Delirium Observation Screening scale is 3 or higher. The Delirium Observation Screening scale ranges from 0 to 39, with higher scores indicating a higher chance of delirium.
30-day incidence of surgical site infections (for surgical patients) | 30 days after admission
  30-day incidence of surgical site infections, as assessed by physicians from the department where patient is admitted during hospitalization. If the patient obtained a surgical site infection after discharge, incidence was assessed in the outpatient clinic by a physician from the department where patient was admitted.
Objective sleep substudy: Sleep efficiency (objectively measured) during admission | Second night of admission (medical patients) and first postoperative night on surgical ward (for surgical patients)
  Objective sleep quality will be measured by the Dreem-3 headband, using electro-encephalography (EEG) to differentiate between wakefulness, Rapid-Eye-Movement (REM) sleep and non-REM N1, N2 and N3 sleep. The primary outcome measure will be sleep efficiency (time slept divided by time in bed spent trying to sleep), compared for patients on intervention and control departments.
Objective sleep substudy: Differences in objective sleep measures of sleep-wake timing during admission | The first night until the seventh night of admission; if the patient is discharged before 7 nights of admission, all nights of admission will be analyzed
  Sleep-wake timing will be assessed by the Dreem-3 headband, using electro-encephalography (EEG) to differentiate between wakefulness, Rapid-Eye-Movement (REM) sleep and non-REM N1, N2 and N3 sleep, and the Withings Sleep Analyzer, differentiating between wakefulness, REM- and light and deep sleep. Changes in sleep-wake timing (i.e. midpoint of sleep, sleep on- and offset time, sleep duration, sleep latency & inertia) will be compared for patients on intervention and control departments.
Objective sleep substudy: Night-to-night changes in objective sleep measures during admission | The first night until the seventh night of admission; if the patient is discharged before seven nights of admission, all nights of admission will be analyzed
  Objective sleep quality will be measured by the Dreem-3 headband, using electro-encephalography (EEG) to differentiate between wakefulness, Rapid-Eye-Movement (REM) sleep and non-REM N1, N2 and N3 sleep, and the WIthings Sleep Analyzer, differentiating between wakefulness, REM- and light and deep sleep. The amount of time in each of these stages and their distribution, as well as total sleep time, will be compared for patients on intervention and control departments.
Objective sleep substudy: Difference between objective and subjective sleep measures during admission | The first night until the seventh night of admission; if the patient is discharged before seven nights of admission, all nights of admission will be analyzed)
  Objective sleep quality will be measured by the Dreem-3 headband, using electro-encephalography (EEG) to differentiate between wakefulness, Rapid-Eye-Movement (REM) sleep and non-REM N1, N2 and N3 sleep, and the WIthings Sleep Analyzer, differentiating between wakefulness, REM- and light and deep sleep. Subjective sleep quality will be measured by the Richard Campbell Sleep Questionnaire, with five questions with a visual analogue scale with scores from 0 to 100, with higher scores indicating better sleep quality. Subjective sleep quantity will be measured with the Consensus Sleep Diary, with questions on sleep-wake timing. Objective and subjective sleep measures will be compared.
Objective sleep substudy: Quality of recovery after surgery and objective sleep quality/timing | First and third day after surgery (surgical patients)
  The association between quality of recovery, as measured by the Quality-of-Recovery 15 item questionnaire (QoR-15), and objective sleep quality and sleep-wake timing (as measured by the Dreem-3 headband, using electro-encephalography (EEG) to differentiate between wakefulness, Rapid-Eye-Movement (REM) sleep and non-REM N1, N2 and N3 sleep, and the Withings Sleep Analyzer, differentiating between wakefulness, REM- and light and deep sleep.). The QoR-15 will be completed twice by patients.
Objective sleep substudy: Correlation 30 day mortality and objective sleep quality/timing | 30 days after admission
  Correlation between 30-day mortality, assessed by checking the medical record retrospectively 30 days after admission and objective sleep quality and sleep-wake timing during admission (as measured by the Dreem-3 headband, using electro-encephalography (EEG) to differentiate between wakefulness, Rapid-Eye-Movement (REM) sleep and non-REM N1, N2 and N3 sleep, and the Withings Sleep Analyzer, differentiating between wakefulness, REM- and light and deep sleep.
Objective sleep substudy: Correlation 30-day incidence of delirium during admission and objective sleep quality/timing | 30 days after admission
  30-day incidence of the clinical diagnosis of delirium during hospitalization, as assessed by a physician during admission. Patients will be assessed for delirium at the request of nursing staff or if the score of the Delirium Observation Screening scale is 3 or higher. The Delirium Observation Screening scale ranges from 0 to 39, with higher scores indicating a higher chance of delirium. Objective sleep quality and sleep-wake timing during admission will be measured by the Dreem-3 headband, using electro-encephalography (EEG) to differentiate between wakefulness, Rapid-Eye-Movement (REM) sleep and non-REM N1, N2 and N3 sleep, and the Withings Sleep Analyzer, differentiating between wakefulness, REM- and light and deep sleep.).
Objective sleep substudy: Correlation 30-day incidence of surgical site infections (for surgical patients) and objective sleep quality/timing | 30 days after admission
  30-day incidence of surgical site infections, as assessed by physicians from the department where patient is admitted during hospitalization. If the patient obtained a surgical site infection after discharge, incidence was assessed in the outpatient clinic by a physician from the department where patient was admitted. Objective sleep quality and sleep-wake timing during admission will be measured by the Dreem-3 headband, using electro-encephalography (EEG) to differentiate between wakefulness, Rapid-Eye-Movement (REM) sleep and non-REM N1, N2 and N3 sleep, and the Withings Sleep Analyzer, differentiating between wakefulness, REM- and light and deep sleep.).

CONTACTS AND LOCATIONS:
Overall Officials: Jeroen j.hermanides@amsterdamumc.nl, PhD, Principal Investigator — Amsterdam UMC; Dirk Jan Stenvers, PhD, Principal Investigator — Amsterdam UMC
Locations (1):
- Amsterdam University Medical Centers, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] de Gans CJ, van den Ende ES, Meewisse AJG, van Zuylen ML, Stenvers DJ, Hermanides J, Nanayakkara PWB. Benzodiazepine receptor agonists in hospitalised patients in the Netherlands: initiation, continuation and discontinuation - a retrospective observational analysis. BMJ Open. 2026 Feb 9;16(2):e112758. doi: 10.1136/bmjopen-2025-112758. PMID 41663167